CLINICAL TRIAL: NCT02461290
Title: Open, Noninterventional, Multicentre Trial of Rituximab in Combination With Chemotherapy (CVP, CHOP or FCM) Chemotherapy in Patients With Follicular Lymphoma
Brief Title: Rituximab Therapy in Follicular Lymphoma in Combination With Chemotherapy - REFLECT 1
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21526
Record Dates: First submitted 2015-05-29; First posted 2015-06-03 (Estimated); Results first posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-08

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Drug Therapy; Rituximab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Combination Therapy: Rituximab 375mg/m2, on day 1 of each cycle of chemotherapy, total of 8 infusions. Chemotherapy according to standard regimens.
  Interventions: Radiation: Chemotherapy; Drug: Rituximab

INTERVENTIONS:
Radiation: Chemotherapy
Drug: Rituximab
  Other Names: MabThera

SUMMARY:
The primary objective is to evaluate the safety profile and tolerability of rituximab in combination with different chemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosed Stage III/IV NHLs
* Grades 1, 2 follicular lymphoma need to be treated
* mCD20 positive
* Have an expected survival of 3 months or more
* ECOG 0-2 grade
* Normal renal function
* ALT less than double normal level

Exclusion Criteria:

* Presence of CNS lymphoma
* Severe infectious disease or organic disease
* Having another malignant tumor
* Pregnant or breast-feeding female
* Organic heart disease, heart failure, II or higher grade AV bundle block.
* Subject is allergic to Rituximab
* Known HIV infection or chronic HBV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with follicular lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2008-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Serbia (5):
  - Belgrade
  - Kamenitz
  - Kragujevac
  - Niš
  - Novi Sad

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab + Chemotherapy: Participants with Stage III or IV, previously untreated follicular lymphoma (FL) received rituximab in combination with chemotherapy, which was prescribed in accordance with local labeling and standard practice at the study site. Chemotherapy regimens included cyclophosphamide, vincristine, and prednisone (CVP); cyclophosphamide, doxorubin, vincristine, and predisone (CHOP); or fludarabine, cyclophosphamide, and mitoxantrone (FCM). Rituximab was administered as 375 milligrams per meter-squared (mg/m^2) via intravenous (IV) infusion on Day 1 of each 21-day cycle for 8 cycles of induction therapy. Because the study was noninterventional, the rituximab regimen was also at the discretion of the prescribing physician.
Period: Overall Study
Arm/Group | Rituximab + Chemotherapy
Started | 99
Completed | 89
Not Completed | 10
Not completed — Withdrawn for Inadequate Clinical Stage | 7
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All participants enrolled into the study.
Groups:
- Rituximab + Chemotherapy: Participants with Stage III or IV, previously untreated FL received rituximab in combination with chemotherapy, which was prescribed in accordance with local labeling and standard practice at the study site. Chemotherapy regimens included CVP, CHOP, or FCM. Rituximab was administered as 375 mg/m^2 via IV infusion on Day 1 of each 21-day cycle for 8 cycles of induction therapy. Because the study was noninterventional, the rituximab regimen was also at the discretion of the prescribing physician.
Arm/Group | Rituximab + Chemotherapy
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event (AE), Serious AE, or Death Related to AE
Description: The safety and tolerability of rituximab was evaluated by collection of AEs, including clinically significant abnormalities and changes in laboratory data. An AE was defined as any untoward medical occurrence in a study participant regardless of the suspected cause. Serious AEs were those which, at any dose, met one or more of the following criteria: resulted in fatality, were life-threatening, necessitated new or prolonged existing hospitalization, produced persistent or significant disability, resulted in a congenital anomaly or birth defect, were considered medically significant, or required intervention to prevent any of the aforementioned outcomes. Those specific serious AEs which resulted in fatality were also reported separately.
Time Frame: Up to 3 years (at Screening, Baseline, end of induction therapy, and in accordance with routine practice)
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | Rituximab + Chemotherapy
Number analyzed (Participants) | 99
participants
  Any AE | 34
  Serious AE | 10
  Death related to AE | 7

2. Secondary Outcome: Percentage of Participants With Complete Remission (CR) or Partial Remission (PR) According to International Working Group Response Criteria for Non-Hodgkin's Lymphoma (NHL)
Description: Tumor response was evaluated according to criteria published by Cheson et al (1999). According to consensus recommendations, CR was defined as disappearance of all clinical/radiographic evidence of disease, regression of lymph nodes to normal size, absence of splenomegaly, and absence of bone marrow involvement. PR was defined as greater than or equal to (≥) 50 percent (%) decrease in sum of the products of greatest diameters (SPD) of the six largest dominant lymph nodes, no increase in size of other nodes, no increase in liver or spleen volume, a ≥50% decrease in SPD of hepatic and splenic nodules, absence of other organ involvement, and no new sites of disease. The percentage of participants achieving CR or PR was calculated as [number of participants meeting the above criteria divided by the number analyzed] multiplied by 100.
Time Frame: Up to 18 months (at Screening, Baseline, end of induction therapy, and in accordance with routine practice)
Population: Data Analysis Population: All enrolled participants who provided complete and evaluable outcome data.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Chemotherapy
Number analyzed (Participants) | 86
percentage of participants | 73.2

3. Secondary Outcome: Percentage of Participants With CR According to International Working Group Response Criteria for NHL
Description: Tumor response was evaluated according to criteria published by Cheson et al (1999). According to consensus recommendations, CR was defined as disappearance of all clinical/radiographic evidence of disease, regression of lymph nodes to normal size, absence of splenomegaly, and absence of bone marrow involvement. The percentage of participants achieving CR was calculated as [number of participants meeting the above criteria divided by the number analyzed] multiplied by 100.
Time Frame: Up to 18 months (at Screening, Baseline, end of induction therapy, and in accordance with routine practice)
Population: Data Analysis Population.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Chemotherapy
Number analyzed (Participants) | 86
percentage of participants | 61.6

4. Secondary Outcome: Percentage of Participants Alive at 1, 2, and 3 Years
Description: Participants were followed for survival for up to 3 years. The overall survival rate at 1, 2, and 3 years was calculated as [number of participants alive divided by the number analyzed] multiplied by 100.
Time Frame: At 1, 2, and 3 years
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Chemotherapy
Number analyzed (Participants) | 99
percentage of participants
  At 1 year | 94.2
  At 2 years | 92.6
  At 3 years | 92.6

ADVERSE EVENTS:
Time Frame: Up to 18 months (at Screening, Baseline, end of induction therapy, and in accordance with routine practice)
Description: ITT Population.
Arm/Group | Rituximab + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 10/99
Other Adverse Events (participants affected / at risk) | 24/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Chemotherapy (N=99)
Encephalitis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Chemotherapy (N=99)
Respiratory tract infection (Infections and infestations) | 3
Herpes simplex (Infections and infestations) | 1
Neutropenia (Blood and lymphatic system disorders) | 17
Pancytopenia (Blood and lymphatic system disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 1
Leucopenia (Blood and lymphatic system disorders) | 12
Hypersensitivity (Immune system disorders) | 4
Immunodeficiency (Immune system disorders) | 1
Hypogammaglobulinaemia (Immune system disorders) | 1
Paresthesia (Nervous system disorders) | 6
Urticaria (Skin and subcutaneous tissue disorders) | 6
Choking (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Hepatic lesion (Hepatobiliary disorders) | 1
Chills (General disorders) | 9
Pyrexia (General disorders) | 13
Infusion related reaction (Injury, poisoning and procedural complications) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.